CLINICAL TRIAL: NCT05377203
Title: Initial Treatment With a Single Capsule Containing Quadruple Combination of Half Doses of Blood Pressure Medicines Versus Standard Dose Dual Therapy in Patients With Hypertension: A Single-center, Randomized, Double-blind, Crossover Trial
Brief Title: Low-dose Quadruple Combination Therapy in Patients With Hypertension
Acronym: QUADUAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R22023; MR-43-23-020339 (Registry Identifier: Medical Research Registration & Information System of China)
Record Dates: First submitted 2022-05-06; First posted 2022-05-17 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Hypertension; Arterial Hypertension
Keywords: hypertension; combination therapy; low dose; randomized controlled trial; crossover design
MeSH Terms: conditions — Hypertension | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: 2×2 crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Persons except who make masking plan and conduct medicine coding, are all masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Quadruple combination of half doses therapy for 4 weeks→Wash out for 2 weeks →Dual combination of standard dose therapy for 4 weeks.
  Interventions: Drug: Quadruple combination of half doses therapy→Dual combination of standard dose therapy
- Group B (Experimental): Dual combination of standard dose therapy for 4 weeks→Wash out for 2 weeks →Quadruple combination of half doses therapy for 4 weeks.
  Interventions: Drug: Dual combination of standard dose therapy→ Quadruple combination of half doses therapy

INTERVENTIONS:
Drug: Quadruple combination of half doses therapy→Dual combination of standard dose therapy — Quadruple combination of half doses therapy: a single capsule containing quadruple combination of half doses of blood pressure medicines (amlodipine besylate tablet 2.5mg, amlodipine besylate tablet simulator 2.5mg, irbesartan tablets 75mg, irbesartan tablets simulator 75mg, metoprolol succinate sustained-release tablets 23.75mg, indapamide tablets 1.25mg), take orally, one capsule once a day.
  Dual combination of standard dose therapy: a single capsule containing dual combination of standard dose of blood pressure medicines (amlodipine besylate tablets 2.5mg×2, irbesartan tablets 75mg×2, metoprolol succinate sustained-release tablets simulator 23.75mg, indapamide tablets simulator 1.25mg), take orally, one capsule once a day.
  Arms: Group A
Drug: Dual combination of standard dose therapy→ Quadruple combination of half doses therapy — Dual combination of standard dose therapy: a single capsule containing dual combination of standard dose of blood pressure medicines (amlodipine besylate tablets 2.5mg×2, irbesartan tablets 75mg×2, metoprolol succinate sustained-release tablets simulator 23.75mg, indapamide tablets simulator 1.25mg), take orally, one capsule once a day.
  Quadruple combination of half doses therapy: a single capsule containing quadruple combination of half doses of blood pressure medicines (amlodipine besylate tablet 2.5mg, amlodipine besylate tablet simulator 2.5mg, irbesartan tablets 75mg, irbesartan tablets simulator 75mg, metoprolol succinate sustained-release tablets 23.75mg, indapamide tablets 1.25mg), take orally, one capsule once a day.
  Arms: Group B

SUMMARY:
This study aims to compare the antihypertensive effect of initial treatment with a single capsule containing quadruple combination of half-dose of blood pressure medicines or standard dose dual combination in patients with hypertension.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, crossover trial, planning to enroll 90 patients with grade 1 and 2 hypertension in the Third Xiangya Hospital of Central South University. The participants will be divided into two groups randomly and treated with half-dose quadruple antihypertensive therapy (irbesartan 75mg+ metoprolol 23.75mg+ amlodipine 2.5mg+ indapamide 1.25mg) or with full-dose dual antihypertensive therapy (irbesartan 150mg+ amlodipine 5mg) for four weeks. After washing out with placebo for two weeks, the participants of the two groups will exchange their medication and be treated for another four weeks. The changes of blood pressure (including 24-hour ambulatory blood pressure, office blood pressure, and home blood pressure) and related adverse effects of the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, < 80 years old；
* Have never taken antihypertensive medications or have not taken antihypertensive medications in the past 1 month；
* Patients with hypertension (meet the following two parameters to avoid white coat hypertension):a. Office Blood Pressure: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg measured 3 times on different days;b. ABPM: average blood pressure of 24h ≥130/80 mmHg; Or average blood pressure of daytime ≥135/85 mmHg; Or average blood pressure of night ≥120/70 mmHg;
* Participate voluntarily and sign written informed consent.

Exclusion Criteria:

* Confirmed or highly suspected secondary hypertension, such as primary aldosteronism, Cushing's syndrome, pheochromocytoma or paraganglioma, aortic constriction, renal arterial stenosis, renal hypertension, hyperthyroidism, etc.;
* Severe hypertension: systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg in the consulting room or hypertensive emergency or urgency at the time of visit;
* Differences in blood pressure of both upper limbs ≥20/10mmHg;
* Allergic to irbesartan, metoprolol, amlodipine, indapamide and sulfonamides;
* Cannot swallow tablets;
* Pregnant and lactating women;
* Possible reproductive needs during the trial;
* Uncorrected electrolyte disorder (serum potassium > 5.5mmol/L or < 3.5mmol/L, serum sodium < 135mmol/L);
* Severe organ dysfunction, including impaired renal function (GFR < 60mL /min/1.73m^2), impaired liver function (aspartate aminotransferase or alanine aminotransferase ≥ 3 times the upper limit of normal), NYHF classification class IV for cardiac function;
* Comorbidities lead to inaccurate blood pressure measurement, such as arrhythmia, etc.;
* Comorbidities result in the prohibition or caution of the experimental drugs, such as: aortic stenosis, mitral valve stenosis, hypertrophic obstructive cardiomyopathy, bilateral renal artery stenosis or renal artery stenosis with solitary kidney, gout, hyperuricemia (serum uric acid >420μmol/L in men or 360μmol/L in women), acute coronary syndrome, sick sinus syndrome, degree II-III of atrioventricular block, severe peripheral vascular disease with high risk of gangrene, history or family history of angioedema;
* Comorbidities affect the absorption, distribution, metabolism and excretion of the experimental drugs such as: gastrointestinal resection, gastrointestinal bypass surgery, sympathetic nerve resection or other operations, active inflammatory bowel disease, malignant tumors undergoing or planning to undergo radiotherapy or chemotherapy or targeted therapy, etc.;
* Medications in use or about to be used may lead to the prohibition or caution of experimental drugs: such as ACEI, Aliskiren, lithium agent, etc.;
* Medications in use or about to be used will interfere the results of this study, such as: hormones, Sacubitril valsartan and spironolactone for patients with chronic heart failure, Dapagliflozin and Liraglutide for patients with diabetes, and long-term medication for patients with chronic coronary heart disease, etc.;
* Not appropriate for antihypertensive therapies of this trial evaluated by physician;
* Participating in other clinical research that may affect the conduct of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Mean systolic blood pressure of 24-hour | Four weeks
  The reduction of mean systolic blood pressure of 24-hour in Ambulatory Blood Pressure Monitoring (ABPM) after 4 weeks of medication (from baseline).

SECONDARY OUTCOMES:
Mean systolic blood pressure of daytime and night | Four weeks
  The reduction of mean systolic blood pressure of daytime and night in ABPM after 4 weeks of medication (from baseline).
Mean diastolic blood pressure of 24-hour, daytime and night | Four weeks
  The reduction of mean diastolic blood pressure of 24-hour, daytime and night in ABPM after 4 weeks of medication (from baseline).
Morning blood pressure surge | Four weeks
  The change of morning blood pressure surge in ABPM after 4 weeks of medication (from baseline).
Office blood pressure | Four weeks
  The reduction of office blood pressure after 4 weeks of medication (from baseline).
Home blood pressure | Four weeks
  The reduction of home blood pressure after 4 weeks of medication (from baseline).
Heart rate | Four weeks
  The change in heart rate after 4 weeks of medication (from baseline).
Controlled rate of blood pressure | Four weeks
  Controlled rate of blood pressure after 4 weeks of medication (from baseline).

OTHER OUTCOMES:
Percentage of participants with severe adverse events (SAE) | Four weeks
  Percentage of participants with any SAE according to Good Clinical Practice definition.
Percentage of participants with side effects | Four weeks
  Percentage of participants with occurrence of any potentially relevant side effect (pre-specified as in study protocol).
Rate of relevant side effects | Four weeks
  Rate of relevant side effects (pre-specified as in study protocol) at the participant level.
Mean change in serum potassium | Four weeks
  Mean change (from baseline) in serum potassium after 4 weeks of medication.
Mean change in serum sodium | Four weeks
  Mean change (from baseline) in serum sodium after 4 weeks of medication.
Mean change in blood urea nitrogen | Four weeks
  Mean change (from baseline) in blood urea nitrogen after 4 weeks of medication.
Mean change in serum creatinine | Four weeks
  Mean change (from baseline) in serum creatinine after 4 weeks of medication.
Mean change in serum uric acid | Four weeks
  Mean change (from baseline) in serum uric acid after 4 weeks of medication.
Mean change in serum glutamic-oxalacetic transaminase | Four weeks
  Mean change (from baseline) in serum glutamic-oxalacetic transaminase after 4 weeks of medication.
Mean change in serum glutamic-pyruvic transaminase | Four weeks
  Mean change (from baseline) in serum glutamic-pyruvic transaminase after 4 weeks of medication.
Mean change in serum bilirubin | Four weeks
  Mean change (from baseline) in serum bilirubin (total and direct bilirubin) after 4 weeks of medication.
Mean change in blood glucose | Four weeks
  Mean change (from baseline) in blood glucose after 4 weeks of medication.
Mean change in urinary protein | Four weeks
  Mean change (from baseline) in urinary protein (-, +, ++, +++) after 4 weeks of medication.
Change in electrocardiogram QT Interval | Four weeks
  Change (from baseline) in electrocardiogram QT Interval after 4 weeks of medication.

CONTACTS AND LOCATIONS:
Overall Officials: Weihong Jiang, Doctor, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and clinical study report will be shared by publishing way.
Supporting Information: Study Protocol, CSR
Time Frame: When study protocol and clinical study report are accepted to publish, they will be available.

REFERENCES:
- [Background] Joint Committee for Guideline Revision. 2018 Chinese Guidelines for Prevention and Treatment of Hypertension-A report of the Revision Committee of Chinese Guidelines for Prevention and Treatment of Hypertension. J Geriatr Cardiol. 2019 Mar;16(3):182-241. doi: 10.11909/j.issn.1671-5411.2019.03.014. No abstract available. PMID 31080465
- [Background] Unger T, Borghi C, Charchar F, Khan NA, Poulter NR, Prabhakaran D, Ramirez A, Schlaich M, Stergiou GS, Tomaszewski M, Wainford RD, Williams B, Schutte AE. 2020 International Society of Hypertension Global Hypertension Practice Guidelines. Hypertension. 2020 Jun;75(6):1334-1357. doi: 10.1161/HYPERTENSIONAHA.120.15026. Epub 2020 May 6. No abstract available. PMID 32370572
- [Background] Lu J, Lu Y, Wang X, Li X, Linderman GC, Wu C, Cheng X, Mu L, Zhang H, Liu J, Su M, Zhao H, Spatz ES, Spertus JA, Masoudi FA, Krumholz HM, Jiang L. Prevalence, awareness, treatment, and control of hypertension in China: data from 1.7 million adults in a population-based screening study (China PEACE Million Persons Project). Lancet. 2017 Dec 9;390(10112):2549-2558. doi: 10.1016/S0140-6736(17)32478-9. Epub 2017 Nov 5. PMID 29102084
- [Background] Chow CK, Gupta R. Blood pressure control: a challenge to global health systems. Lancet. 2019 Aug 24;394(10199):613-615. doi: 10.1016/S0140-6736(19)31293-0. Epub 2019 Jul 18. No abstract available. PMID 31327567
- [Background] An J, Luong T, Qian L, Wei R, Liu R, Muntner P, Brettler J, Jaffe MG, Moran AE, Reynolds K. Treatment Patterns and Blood Pressure Control With Initiation of Combination Versus Monotherapy Antihypertensive Regimens. Hypertension. 2021 Jan;77(1):103-113. doi: 10.1161/HYPERTENSIONAHA.120.15462. Epub 2020 Nov 16. PMID 33190560
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Derived] Zhao X, Liu T, Yang Q, Yang G, Li X, Tang X, Li J, Liang Z, Li A, Zeng L, Wen J, Wang X, Peng L, Wang W, Cai J, Chen Y, Huang M, Li R, Fu R, Zhao L, Li X, Jiang W. Initial treatment with a single capsule containing half-dose quadruple therapy vs standard-dose dual therapy in hypertensive patients (QUADUAL): a randomized, blinded, crossover trial. BMC Med. 2025 Jan 29;23(1):56. doi: 10.1186/s12916-025-03892-8. PMID 39881316
- [Derived] Zhao X, Li X, Liu T, Yang G, Chen Y, Huang M, Zhao L, Li X, Jiang W. Initial treatment with a single capsule containing half-dose quadruple therapy versus standard-dose dual therapy in hypertensive patients (QUADUAL): statistical analysis plan for a randomized, blinded, crossover trial. Trials. 2024 Jan 13;25(1):45. doi: 10.1186/s13063-023-07803-1. PMID 38218924
- [Derived] Zhao X, Chen Y, Yang G, Li X, Tang X, Yang Q, Peng L, Li J, Liang Z, Li A, Wang W, Huang M, Liu T, Li X, Jiang W. Initial treatment with a single capsule containing half-dose quadruple therapy vs standard-dose dual therapy in hypertensive patients (QUADUAL): Study protocol for a randomized, blinded, crossover trial. Am Heart J. 2023 Oct;264:10-19. doi: 10.1016/j.ahj.2023.05.019. Epub 2023 Jun 4. PMID 37276913
- Available data/document: Study Protocol: PMID: 37276913 — https://www.ncbi.nlm.nih.gov/pubmed/37276913